CLINICAL TRIAL: NCT06614764
Title: Effect of Andiroba on Control of Post-whitening Tooth Sensitivity: a Randomized Clinical Trial
Brief Title: Effect of Andiroba on Control of Post-whitening Tooth Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Professor of the Graduate Program in Dentistry at the Federal University of Pará, Universidade Federal do Para
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 81021724.2.0000.0018
Record Dates: First submitted 2024-09-20; First posted 2024-09-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-09

CONDITIONS: Tooth Bleaching; Pain; Dentin Desensitizing Agents
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PG- Placebo gel (Placebo Comparator): The PG group received the application of placebo gel for post tooth bleaching sensitivity.
  Interventions: Other: PG (Placebo Gel)
- GKF2- Potassium nitrate (Active Comparator): The KF2 group received the application of potassium nitrate for post tooth bleaching sensitivity.
  Interventions: Other: KF2G (Potassium nitrate gel)
- AG- Andiroba Gel (Experimental): The AG group received the application of experimental gel of andiroba (Carapa guianensis) for post tooth bleaching sensitivity.
  Interventions: Other: AG (experimental Andiroba Gel)

INTERVENTIONS:
Other: AG (experimental Andiroba Gel) — Prior to bleaching treatment with 35% hydrogen peroxide, the dental elements of the AG received application of the experimental desensitizing gel on the buccal surfaces of the central incisors, lateral incisors, canines and upper and lower premolars, with a rubber cup in an active way, for 10 minutes.
  Arms: AG- Andiroba Gel
Other: KF2G (Potassium nitrate gel) — Prior to bleaching treatment with 35% hydrogen peroxide, the dental elements of the KF2G received application of the potassium nitrate gel on the buccal surfaces of the central incisors, lateral incisors, canines and upper and lower premolars, with a rubber cup in an active way, for 10 minutes.
  Arms: GKF2- Potassium nitrate
Other: PG (Placebo Gel) — Prior to bleaching treatment with 35% hydrogen peroxide, the PG group received the application of a placebo gel (without active ingredient), under the same conditions described for the experimental gel.
  Arms: PG- Placebo gel

SUMMARY:
This randomized clinical trial will evaluate the effect of an experimental gel containing andiroba oil (Carapa guianensis) in reducing postoperative tooth sensitivity caused by bleaching with 35% hydrogen peroxide. Volunteers in this study will be randomized into 3 different groups - PG (placebo gel), KF2G (potassium nitrate gel) and AG (andiroba gel). Groups KF2G and AG will receive treatment with potassium nitrate desensitizing gel and the experimental andiroba gel, respectively. This will be applied to the buccal surfaces of the central incisors, lateral incisors, canines and upper and lower premolars, with a rubber cup in an active manner, for 10 minutes. Group GP will receive the application of a placebo gel (without active ingredient), under the same conditions described for the other groups. Subsequently, all groups will undergo in-office bleaching treatment with 35% hydrogen peroxide. Post-bleaching sensitivity will be collected using a form consisting of the visual analogue scale (VAS). Color measurement will be performed with a spectrophotometer at two times: baseline (T0) and one week after the 3rd bleaching session (T1).

DETAILED DESCRIPTION:
All groups will undergo in-office whitening treatment, carried out in 3 sessions with a 7-day interval, according to the steps described below:

Prophylaxis; Application of gingival barrier; Application of desensitizing agent or placebo, according to the established groups; Handling of the whitening material following the manufacturer's instructions: application of Whiteness HP 35% whitening gel for 15 minutes each, totaling 45 minutes; Final removal of the whitening gel and gingival barrier, followed by rinsing with water.

The application of the desensitizing agent or its placebo will follow this sequence:

Relative isolation with cotton rolls; Active application of the product on the buccal surfaces of all teeth using a rubber cup for 10 minutes; Rinsing with water.

ELIGIBILITY:
Inclusion Criteria:

* good oral hygiene
* absence of active caries lesions
* never having undergone previous whitening therapy
* not present dental hypersensitivity
* don't be a smoker
* not be pregnant
* present at least 28 teeth in the oral cavity.

Exclusion Criteria:

* volunteers who were under orthodontic treatment,
* presence of periodontal disease
* dental cracks or fractures
* restorations and prostheses on anterior teeth
* extensive molar restorations
* gastroesophageal disorders
* severe internal dental darkening
* presence of dentinal exposure in anterior and / or posterior teeth.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Post-whitening sensitivity assessment | Period: 21 days
  To assess post-operative sensitivity, patients will be instructed to fill out a form to record daily tooth sensitivity during the 21 days of treatment, based on their individual perception of pain. This form will be handed out at each whitening session and returned to the researcher at the following session, that is, always one week after each whitening session. The assessment form will consist of a visual analogue scale (VAS). This scale consists of a 10 cm horizontal line with scores of 0 and 10 at its ends, where 0 means no sensitivity and 10 means severe tooth sensitivity. The patient will be instructed to draw a vertical line along the horizontal line of the scale, recording the intensity of tooth sensitivity per day. So that the distance in millimeters from the zero end can later be measured with the aid of a millimeter ruler, thus obtaining the patient's pain intensity level.

SECONDARY OUTCOMES:
Color evaluation | Baseline (Ti) and one week after the 3rd whitening session (Tf).
  The VITA Easyshade spectrophotometer (VITA Zahnfabrik, Bad Säckingen, Germany) will be used to measure the color, where the area of dental correspondence to be evaluated will be the middle third of the vestibular surface of the upper canines. To standardize the color readings, silicone matrices will be made, where the impression will be extended from canine to canine. A window will be created on the vestibular surface of each canine of the silicone guide using a metal device with a radius of 6 mm, corresponding to the diameter of the spectrophotometer tip. Thus, the tip of the device will be inserted into the silicone guide to obtain the color parameters. Subsequently, the color difference between the baseline (T0) and one week after the 3rd bleaching session (T1) will be calculated using the CIEDE2000 formulas (ΔE00).

CONTACTS AND LOCATIONS:
Overall Officials: Cecy M Silva, doctor, Principal Investigator — Universidade federal do Pará
Locations (1):
- UFPA, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No